CLINICAL TRIAL: NCT00486382
Title: A Phase 1, Open-Label, Dose Escalating Study to Evaluate the Safety, Tolerability, and Immunogenicity of the LEISH-111F + MPL-SE Vaccine (Recombinant Three-Antigen Leishmania Polyprotein With Adjuvant MPL-SE) in Healthy Adults In India
Brief Title: Open-Label Safety Study of Three-Antigen Leishmania Polyprotein With Adjuvant MPL-SE in Healthy Adults in India
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRI-LVVPX-104
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Visceral Leishmaniasis; Post-kala-azar Dermal Leishmaniasis
Keywords: visceral leishmaniasis; vaccine
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): Biological/Vaccine: Leish-111f + MPL-SE Adjuvant
  Interventions: Biological: Leish-111f + MPL-SE Adjuvant
- Medium dose (Experimental): Biological/Vaccine: Leish-111f + MPL-SE Adjuvant
  Interventions: Biological: Leish-111f + MPL-SE Adjuvant
- High dose (Experimental): Biological/Vaccine: Leish-111f + MPL-SE Adjuvant
  Interventions: Biological: Leish-111f + MPL-SE Adjuvant

INTERVENTIONS:
Biological: Leish-111f + MPL-SE Adjuvant

SUMMARY:
The purpose of this study is to determine if a vaccine (called Leish-111f + MPL-SE) is safe and whether it can or cannot produce a protective response against visceral leishmaniasis when injected to healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety, tolerability, and immunogenicity of an investigational vaccine being developed for immunotherapy of visceral leishmaniasis (VL) and post kala-azar dermal leishmaniasis (PKDL). The vaccine, identified as Leish-111f + MPL-SE, consists of a recombinant three-antigen Leishmania polyprotein (Leish-111f) together with adjuvant MPL-SE.

The primary objective is to evaluate the safety and tolerability of the Leish-111f + MPL-SE vaccine given as three subcutaneous injections every 28 days at each of three dose levels of the Leish-111f protein (5 μg, 10 μg, or 20 μg) together with MPL-SE adjuvant (25 μg) in healthy adults.

The secondary objective is to assess the immunogenicity of the vaccine by evaluating T-cell and antibody response to the Leish-111f protein of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years and < 55 years of age.
* Must be in good general health as confirmed by a medical history and physical exam.
* DAT titer must be <1:400 and rK39 serology negative (for inclusion in the DAT-negative group) or DAT titer ≥1:1600 (for inclusion in the DAT-positive group).
* The following laboratory blood tests must have values within the normal ranges at screening (Appendix 4): sodium, potassium, urea, ALT, AST, total bilirubin, creatinine, alkaline phosphatase, glucose, hemoglobin, total WBC count and platelet count.
* The following serology tests must be negative at screening: HIV 1/2, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. All subjects will receive HIV related counseling prior to testing. Subjects with positive HIV test results will receive counseling at the University and will be referred to the national AIDS control program for treatment if appropriate.
* Subjects must give written informed consent, be willing and able to attend all required visits, have a permanent address, and be reachable by study site personnel.
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening, a negative urine pregnancy test within 24 hours before study injection, must not be breast-feeding, and are required to use adequate contraception through Day 84 of the study. These precautions are necessary due to unknown effects that Leish-111f + MPL-SE might have in a fetus or newborn infant.

Exclusion Criteria:

* Previous exposure to Leishmania vaccines or experimental products containing MPL-SE.
* Participation in another experimental protocol or receipt of any investigational products within 30 days prior to the first administration of study injection.
* Known use of injected or oral corticosteroids within 6 weeks prior to the first administration of study injection.
* History of autoimmune disease or other causes of immunosuppressive states.
* History or evidence of any acute or chronic illness that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or the immunogenicity of the vaccine. (Potential subjects presenting with concomitant illness will be referred for clinical care.)
* History of use of any medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or the immunogenicity of the vaccine.
* History of significant psychiatric illness.
* Known to be a current drug or alcohol abuser.
* Subjects with a history of previous anaphylaxis, severe allergic reaction to vaccines or unknown allergens, or allergic reaction to eggs.
* History of chronic headaches or migraine.
* Subjects who are unlikely to cooperate with the requirements of the study protocol.
* Subjects who are not permanent residents or who are planning to move to another town/city.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Injection site reactions | For 7 days following each injection.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Banaras Hindu University; Franco M Piazza, MD, MPh, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India